CLINICAL TRIAL: NCT02632214
Title: Plasticity and Cross-modal Interactions for Oral Communication in Profoundly Deaf Adults
Brief Title: Plasticity and Cross-modal Interactions in Profoundly Deaf Adults
Acronym: PLASMODY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Centre National de la Recherche Scientifique, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Basic Science
Other Study IDs: 2014-A00088-39
Record Dates: First submitted 2015-08-11; First posted 2015-12-16 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Deafness; Perception, Bilateral
Keywords: Face processing; asymmetry; deaf; fMRI
MeSH Terms: conditions — Deafness

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Deaf (Experimental): Group of early profound deaf participants fMRI measure
  Interventions: Other: fMRI measure
- Hearing signers (Experimental): Group of hearing signer controls fMRI measure
  Interventions: Other: fMRI measure
- Hearing non signers (Sham Comparator): Group of hearing non signer controls fMRI measure
  Interventions: Other: fMRI measure

INTERVENTIONS:
Other: fMRI measure

SUMMARY:
The aim of this study is to evaluate cerebral asymmetry for face processing in a group of profoundly deaf participants and a group of hearing controls by the mean of fMRI measure. To this end, we present chimeric faces (faces split into different halves), entire faces, or faces presented in divided visual field, and subjects perform a gender categorization task while lying in a fMRI scanner.

It is expected to find a reduced cerebral asymmetry in the Fusiform Face Area in deaf in comparison with hearing participants.

DETAILED DESCRIPTION:
A rightward asymmetry during face processing is well documented in hearing participants, in particular in the Fusiform Face Area, a cortical area underlying face processing. This rightward asymmetry seems to be very robust, present even with inverted faces or line drawings, and is already present at five years of age. If the brain asymmetry for face processing emerges during development, early deprivation or dramatic differences the infant's experience with the world should affect it. For example, infants treated for bilateral congenital cataracts after 7 weeks of age, who are deprived of patterned visual input for this duration, fail to develop some of the aspects associated with typical adult levels of face recognition. Non visual early deprivation can also affect the development of visual abilities. Several studies showed that deaf participants could detect targets at larger eccentricities, thus indicating larger visual field . Furthermore, better abilities have been found in deaf participants for the detection of motion, in particular in the visual periphery . Higher-level visual abilities have also been shown to be modified by early deafness, such as visual imagery (image generation, or rotation) or the processing of faces . Using the Benton Test of Facial Recognition, a previous study tested the recognition of individual faces in deaf participants. They obtained better scores than hearing non signers, but only in a difficult condition, in which faces were shadowed. This enhanced processing in deaf people could thus concern very particular aspects of face processing; it was found that deaf and normal hearing differed only by the detection of subtle facial features. Investigating configural processing during face perception, it was found an increased dependency on this mode of processing in deaf participants.

If visual processing is affected by early deafness, what about visual asymmetries? Several experimental studies examining hemispheric asymmetry in congenitally deaf individuals found that it differs from the one observed in hearing individuals . Concerning face processing, few studies investigated hemispheric lateralization during the perception of faces in deaf people. When presenting briefly unfamiliar faces in either the left or right visual field and no differences between deaf and hearing participants were found. In a previous experiment, using chimeric faces (faces vertically split into two different parts, ie half male, half female) it was found a reduction of leftward asymmetry for face processing in deaf participants during a gender categorization task.

The aim of the present study is to broaden the knowledge about asymmetry for face processing in deaf people, by evaluating if this reduction of asymmetry observed at the behavioral level results from a reduction of cerebral asymmetry at the level of Fusiform Face Area.

Deaf participants and normal hearing controls will be presented face stimuli, composed of either chimeric male/female and female/male faces, entire faces or entire face presented in divided visual field, to investigate Fusiform Face Area asymmetry in these two groups. Participants will lie in an fMRI scanner, and their cerebral activity will be recorded while they perform a gender categorization task on our face stimuli.

ELIGIBILITY:
Inclusion Criteria:

* Consent Form signed
* Medical exam performed before entering in to the scanner
* age between 18 and 60 years
* Absence of neurological and/or psychiatric troubles
* Normal or corrected vision
* Right handed

For Deaf participants:

* Bilateral hearing loss 80 dB or more
* Hearing loss before 2 years of age
* use of French Sign Language

For Hearing participants - signers:

* Absence of hearing loss
* Use of French sign Language (Bilingual)

For Hearing participants - non signers:

* Absence of hearing loss

Exclusion Criteria:

* Pregnant women, mothers who suckle, minors
* Presence of metal implants (cardiac implants, bone implants, auditory implants...),
* Presence of skin implants: not removable body piercings, tattoos, not removable jewels
* Claustrophobia
* Visual impairment without correction
* Neurological/Psychiatric disorder
* Cardiac or respiratory trouble

For Deaf participants:

* unilateral hearing loss
* cochlear implant

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2014-04; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
cerebral activity (fMRI measure) | Time 0

CONTACTS AND LOCATIONS:
Locations (1):
- plateforme IRMage, Grenoble, France